CLINICAL TRIAL: NCT01170650
Title: A Randomized Double-Blind Phase 3 Trial Comparing EC145 and Pegylated Liposomal Doxorubicin (PLD/Doxil®/Caelyx®) in Combination Versus PLD in Participants With Platinum-Resistant Ovarian Cancer
Brief Title: Study for Women With Platinum Resistant Ovarian Cancer Evaluating EC145 in Combination With Doxil® (PROCEED)
Acronym: PROCEED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB decision
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8109-002; EC-FV-06 (Other: Endocyte)
Record Dates: First submitted 2010-07-07; First posted 2010-07-27 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Cancer
Keywords: cancer; ovarian; platinum-resistant; Phase III; EC145; EC20
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — EC145; liposomal doxorubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): EC145 + Pegylated Liposomal Doxorubicin (PLD)
  Interventions: Drug: EC145; Drug: Pegylated Liposomal Doxorubicin (PLD/Doxil®/Caelyx®); Drug: EC20
- Arm B (Active Comparator): placebo + Pegylated Liposomal Doxorubicin (PLD)
  Interventions: Drug: Pegylated Liposomal Doxorubicin (PLD/Doxil®/Caelyx®); Drug: placebo; Drug: EC20

INTERVENTIONS:
Drug: EC145 — IV bolus on days 1,3,5 and 15,17,19 of a 4-week cycle
  Arms: Arm A
Drug: Pegylated Liposomal Doxorubicin (PLD/Doxil®/Caelyx®) — 50 mg/m2 (calculated on the basis of ideal body weight) every 4 weeks. Dose reductions permitted for toxicity.
  Other Names: Doxil; Caelyx
Drug: placebo — IV bolus on days 1,3,5 and 15,17,19 of a 4-week cycle
  Arms: Arm B
Drug: EC20 — During the screening period participants will receive a single intravenous administration of EC20 prior to SPECT imaging

SUMMARY:
The purpose of this study is to compare progression-free survival (PFS) (based upon investigator assessment using RECIST v1.1) in participants with platinum-resistant ovarian cancer who receive combination therapy with EC145 and pegylated liposomal doxorubicin (EC145+PLD) with that in participants who receive PLD and placebo.

DETAILED DESCRIPTION:
This is a Phase 3 clinical trial to evaluate the efficacy and safety of the combination of EC145 and pegylated liposomal doxorubicin (PLD; available in the United States as Doxil® and outside the United States as Caelyx®) compared to PLD and placebo. Enrollment of 640 patients including approximately 500 that are folate receptor positive is planned.

EC145 is a drug that is specifically designed to enter cancer cells via the folate vitamin receptor (FR) that is not generally found on normal cells. Experimental evidence shows that this target receptor is expressed on virtually all ovarian cancers. Early clinical evidence in a small number of Phase I participants, in a subset of participants in a completed single-arm Phase II study, and interim data from an ongoing randomized Phase 2 study (PRECEDENT) suggests that EC145 may have antitumor effect in women with platinum-resistant ovarian cancer and that EC145 alone and in combination with PLD is generally well-tolerated. This evidence suggests that EC145 may be useful as chemotherapy against platinum-resistant ovarian cancer.

All participants will undergo imaging with the FR-targeting investigational diagnostic agent EC20 during the screening period to assess binding of the imaging agent EC20 to tumors. This non-invasive procedure will provide additional information on the utility of using EC20 imaging to identify subjects with the FR molecular "target" prior to treatment with EC145 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign an approved informed consent form (ICF).
* Participants must be ≥ 18 years of age.
* Participants must have pathology-confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Participants must have primary or secondary platinum-resistant ovarian cancer.
* Participants must have at least a single (RECIST v1.1-defined) measurable lesion.
* For the purpose of obtaining a RECIST v1.1 baseline scan, participants must have a radiological evaluation conducted no more than 28 days prior to beginning study therapy (PLD). NOTE: For participants with a history of CNS metastasis, baseline radiological imaging must include an evaluation of the head.
* Participants must have had prior debulking surgery.
* Participants must have received prior platinum-based chemotherapy for management of primary disease but must not have received more than 2 prior systemic cytotoxic regimens.
* Participants are allowed to have received, but are not required to have received, one additional non-cytotoxic antitumor agent (eg, biologic or cytostatic) for the management of ovarian cancer.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Participants must have recovered (to baseline/stabilization) from prior cytotoxic therapy-associated acute toxicities.
* Participants must have adequate organ function including:

  1. Bone Marrow Reserve:

     1. Absolute neutrophil count (ANC) ≥ 1.5x10^9/L prior to treatment. Participants on maintenance doses of granulocyte colony stimulating factor (G-CSF) are eligible.
     2. Platelets ≥ 100x10^9/L
     3. Hemoglobin ≥ 9 g/dL
     4. Use of supportive care measures (eg, use of white blood cell [WBC] growth factors, antiemetics, epoetin) should follow the ASCO guidelines as listed at www.asco.org. Participants should receive full supportive care, including transfusion of blood as mandated by clinical need; however, transfusions administered for the sole purpose of meeting the study inclusion criteria between the time informed consent is signed and first dose of EC145/placebo/PLD is administered are not allowed.
  2. Hepatic: Total bilirubin level < 1.5 x ULN and ALT, AST, GGT, and alkaline phosphatase levels < 2.5 x ULN.
  3. Renal: Serum creatinine level ≤ 1.5 x ULN or for participants with serum creatinine levels above 1.5 x ULN, creatinine clearance ≥ 50 mL/min/1.73m^2
  4. Cardiac: Left ventricular ejection fraction (LVEF) equal to or greater than the institutional lower limit of normal.

Exclusion Criteria:

* Patients refractory to primary platinum therapy where "refactory" is defined as disease progression within 6 months of first dose of initial platinum-based therapy.
* Diagnosis of "tumor of low-malignant potential".
* Prior exposure to PLD or anthracycline therapy.
* Prior exposure to FR-targeted therapy (eg, EC145, EC0225, EC0489, farletuzumab).
* Prior therapy with vinorelbine (Navelbine®) or vinca-containing compounds.
* Prior abdominal or pelvic radiation therapy or radiation therapy to > 10% of the bone marrow at any time in the past or prior radiation therapy within the past 3 years to the breast/sternum, dermal lesions, head or neck.
* Recent (i.e., ≤ 6 weeks) history of abdominal surgery or peritonitis
* Serious comorbidities (as determined by the investigator) such as, but not limited to, active congestive heart failure or recent myocardial infarction. Patients who require antifolate therapy for the management of comorbid conditions (e.g., rheumatoid arthritis) will be excluded from the trial.
* Pregnant or nursing.
* Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ).
* Symptomatic central nervous system (CNS) metastasis.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation). Use of low dose corticosteroid therapy (e.g., for nausea prophylaxis) is acceptable; however, concomitant tamoxifen therapy is not. Supportive care measures are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2011-04-22; Primary Completion 2015-05-31 (Actual); Study Completion 2015-09-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival based on investigator assessment using RECIST v1.1. | up to 26 months
  Progression is assessed at 6 week intervals through Week 24 and at 8 week intervals thereafter.

SECONDARY OUTCOMES:
Compare overall survival of participants between treatment arms. | Approximately 20 months after last patient randomized
  OS analysis will occur when 384 deaths have occurred.
Incidence of Adverse Events, Serious Adverse Events, and Deaths. | up to 26 months
  Adverse events (as a measure of safety and tolerability) will be assessed at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Binh Nguyen, MD, Study Director — Endocyte

REFERENCES:
- See also: Endocyte website — http://www.endocyte.com